CLINICAL TRIAL: NCT05370807
Title: A Phase-2 Clinical Trial of Regorafenib in Patients With Pretreated Advanced Melanoma - Definition of Two Additional Stratified Patient Cohorts of Regorafenib Plus BRAF-/MEK-inhibitors in Pretreated BRAF V600-mutant Melanoma Patients
Brief Title: A Clinical Trial of Regorafenib in Patients With Pretreated Advanced Melanoma
Acronym: RegoMel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BN-002
Record Dates: First submitted 2022-04-25; First posted 2022-05-12 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-05

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — regorafenib; Tablets

STUDY DESIGN:
Intervention Model Description: 3 cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): Patients take 2 oral tablets of 40mg of Regorafenib daily.
  Interventions: Drug: Regorafenib 40 MG Oral Tablet
- Cohort B (Experimental): Patients take 1 oral tablets of 40mg of Regorafenib daily in combination with BRAF- /MEK- inhibitors dabrafenib/trametinib or encorafenib/binimetinib at the dose they were already taking them.
  Interventions: Drug: Triplet therapy
- Cohort C (Experimental): Patients take 1 oral tablets of 40mg of Regorafenib daily in combination with encorafenib/binimetinib at the standard dose.
  Interventions: Drug: Triplet therapy

INTERVENTIONS:
Drug: Regorafenib 40 MG Oral Tablet — Patients take 2 regorafenib oral tablets of 40 mg daily
  Arms: Cohort A
Drug: Triplet therapy — Regorafenib in combination with BRAF- / MEK- inhibitors
  Arms: Cohort B; Cohort C

SUMMARY:
There are in total 3 cohorts. Cohort A: 16 patients will receive a daily dose of 80mg regorafenib up until progressive disease, unacceptable toxicity or withdrawal of consent. Dose can be escalated intra-patient up to 120 mg if no AE with a grad >1 at 28 days. Patients get a baseline evaluation and have a consultation every 2 weeks for evaluation during treatment. This evaluation consists out of lab tests, PET/CT (not bi-weekly), MRI (not bi-weekly) and physical evaluation.

Primary endpoint is the anti-tumor activity, secondary endpoints are the Overall Survival Rate, Progression Free Survival and the incidence and severity of AE and Health-Related Quality of Life.

Cohort-B: 16 patients who are being treated with BRAF-/MEK- inhibitors will receive additional daily regorafenib in combination with BRAF-/MEK inhibitors. Approved BRAF-/MEK- inhibitor combinations include dabrafenib/trametinib and encorafenib/binimetinib. An interruption of BRAF-/MEK-inhibitors dosing of maximum 4 weeks is allowed between the documentation of progression of disease on this therapy and the initiation of regorafenib study treatment. Dose of regorafenib is 40mg.

Cohort-C: 16 patients in Cohort-C will have interrupted treatment with any BRAF- /MEK - inhibitor combination for at least 12 weeks prior to initiating study therapy with regorafenib. At the time of initiating regorafenib study treatment at 40mg, patients will also resume treatment with encorafenib/binimetinib at its standard dosing regimen.

The first 6 patients enrolled in each Cohort (B, and -C) will be considered as a safety lead-in study population. If two or more serious treatment-related adverse events are observed among the first 6 patients, enrollment will be suspended (if applicable).

The risk/benefit for continuing enrollment will be evaluated and an interim safety report will be provided to the Medical Ethics Committee of the UZ Brussel. If less than two serious treatment-related adverse events are observed, enrollment will be continued without interruption to complete the phase II objective.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Signed written informed consent.
3. Histologically confirmed advanced melanoma that is either stage III (unresectable) or stage IV (metastatic, unresectable)
4. Subjects must have failed prior systemic treatment with immune checkpoint inhibitors, including CTLA-4 blocking immune checkpoint inhibitors (ipilimumab or other experimental anti-CTLA-4 antibodies), and PD-1 blocking immune checkpoint inhibitors (pembrolizumab, nivolumab or other experimental anti-PD-1 antibodies). Progression of disease per RECIST, version 1.1 (Eisenhauer et al. Eur J Cancer 2009) or per immune related response criteria (Wolchok et al, Clin Cancer Res 2009) must have been documented during this prior treatment. Patients with BRAFV600mutant melanoma must have failed treatment with a BRAF-(+/-MEK) inhibitor. Patients who are not able to undergo such treatment will be considered eligible if all other eligibility criteria are fulfilled.
5. The presence of at least one measurable lesion per RECIST, version 1.1 (Eisenhauer et al. Eur J Cancer 2009)
6. Interval between the date of the last administration of prior therapy for melanoma and the date of recruitment:

   1. ≥ 12 weeks following the date of the first administration and ≥ 3 weeks following the date of the last administration of an anti-CTLA-4-, PD-1- or PD-L1 blocking immune checkpoint inhibitor;
   2. ≥ 4 weeks following the date of the last administration of chemotherapy (≥ 6 weeks in case of a nitrosurea or mitomycin C containing regimen);
   3. Cohort-C: ≥ 12 weeks following the date of the last administration of BRAF-/MEK-inhibitors.
7. All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed on Table 1) and non-medical treatments (e.g. surgery and radiation therapy) must be ≤ Grade 1 severity according to the Common Terminology Criteria for Adverse Events version 5 (CTCAE version 5.0; National Cancer Institute (NCI) 2017) at the time of enrollment.
8. The patient must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
9. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to recruitment and agree to use effective contraception throughout the treatment period, and for 16 weeks after the last dose of study treatment.
10. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 14 days prior to administration of the first dose of study treatment, throughout the treatment period, and for 16 weeks after the last dose of study treatment.
11. An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Oken et al, Am J Clin Oncol 1982).
12. Adequate baseline organ function as defined in Table 1.
13. Negative proteinuria on dipstick or 24 hours proteinuria <1000mg.
14. Cohort-B and -C: the melanoma must carry a documented BRAFV600 mutation.
15. Cohort-B: patients should be on treatment with BRAF-/MEK-inhibitors or have interrupted for less than 4 weeks before initiation of the study treatment.
16. Cohort-C: patients should be off BRAF-/MEK-inhibitors for at least 12 weeks before initiation of the study treatment.

Exclusion Criteria:

* 14. Subjects with uveal melanoma. 15. Subjects with clinically active brain metastases (lesions should be stable and have been definitely treated with stereotactic radiation therapy, surgery or gamma knife therapy with no evidence of disease progression prior to enrollment).

  16. Any contra-indication for evaluation by whole body 18F-FDG-PET/CT or MRI of the brain.

  17. History of another malignancy. Exception: subjects who have been disease-free for 3 years, (i.e. subjects with second malignancies that are indolent or definitively treated at least 3 years ago) or subjects with a history of completely resected non-melanoma skin cancer.

  18. Current use of any prohibited medication. 19. Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to recruitment.

  20. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.

  21. Known Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Exception: subjects with laboratory evidence of cleared HBV and HCV infection will be permitted.

  22. Ongoing infection CTCAE v5.0 Grade > 2 requiring systemic therapy. 23. No enzyme inducing anticonvulsants for ≥ 4 weeks prior to recruitment 24. A history or evidence of cardiovascular risk including any of the following:
  1. Current LVEF < LLN
  2. A QT interval corrected for heart rate using the Bazett's formula (QTcB) ≥ 480 msec;
  3. A history or evidence of current clinically significant uncontrolled arrhythmias. Exception: subjects with atrial fibrillation controlled for > 30 days prior to recruitment are eligible.
  4. A history (within 6 months prior to recruitment) of acute coronary syndromes (including myocardial infarction or unstable angina), or coronary angioplasty;
  5. History of deep venous or arterial thrombosis, or CVA the last 6 months
  6. A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines;
  7. Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy;
  8. Patients with intra-cardiac defibrillators or permanent pacemakers;
  9. Abnormal cardiac valve morphology (≥ grade 2; moderate valvular thickening) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study).

     25. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).

     26. Female patients who are nursing. Prior/Concomitant therapy 27. Prior treatment with regorafenib. 28. Cohort-B: 28.1. Patients treated with vemurafenib/cobimetinib 28.2. Patients who are unable to initiate regorafenib within 4 weeks after interruption BRAF-

     /MEK-inhibitor therapy 29. Cohort-C: 29.1. Patients who have not interrupted BRAF-/MEK-inhibitor therapy for at least 12 weeks prior to initiation of study treatment. 30. Patients who received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis. Participants must have recovered from all radiation-related toxicities. A 1-week washout is permitted for palliative radiation (duration of ≤2 weeks of radiotherapy) 31. Patients who have received a live vaccine or live attenuated replication competent vaccine within 32 days prior to the first dose of study treatment. Administration of non-live vaccines are allowed.

     33. Prior transplantation of human cells, tissues and organs (e.g. liver transplant) or candidates for any type of transplantation. 34. Patients on concomitant use of CYP3A4 inducers, strong CYP3A4 inhibitors and strong UGT1A9 inhibitors (e.g. mefenamic acid, diflunisal, and niflumic acid) within 2 weeks prior to start of study treatment. Prior/Concurrent Clinical Study Experience 35. Previous administration of an investigational drug within 28 days, or 5 half-lives (minimum 14 days) before the start of study treatment, whichever is shorter) or concomitant participation in another clinical study with investigational medicinal product(s). Other Exclusions 36. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator. 37. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures. 38. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. 39. Current use of any prohibited medication. 40. Any contra-indication for evaluation by whole body 18F-FDG-PET/CT and/or MRI of the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To measure the anti-tumor acitivity of regorafenib treatment in patients with advanced pretreated melanoma. | Through study completion, an average of 1 year.
  Objective response rate (ORR; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1

SECONDARY OUTCOMES:
To measure the progression-free survival (PFS) of study patients treated with regorafenib | Through study completion, an average of 1 year.
  Progression-free survival (PFS; defined as the time from the date of the first dose administration of regorafenib until the earliest date of documented disease progression [per RECIST v1.1] or death due to any cause)
To measure the overall survival (OS) of study patients treated with regorafenib | Through study completion, an average of 1 year.
  overall survival (OS; defined as the time from the date of the first dose administration of regorafenib until the date of death due to any cause)
Number of AE in study patients | Through study completion, an average of 1 year.
  To count the number of Adverse Events study patients have during the study.
To measure the severity of AE in study patients | Through study completion, an average of 1 year.
  Document the grade of all AE in study patients, expressed in grade 1 Mild, 2 Moderate, 3 Severe, 4 Life-Threatening, 5 Death related to AE
To measure the Health-Related Quality of Life | Through study completion, an average of 1 year.
  There will be 1 questionnaire used to assess the quality of life. The generic health status of the patients will be assessed by means of the EuroQOL-5D-3L (EQ-5D-3L).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussels, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided